CLINICAL TRIAL: NCT04918290
Title: A Randomized Controlled Trial of Tegaderm Vs. Transpore for Eye Protection During Anesthesia
Brief Title: Tegaderm Vs. Transpore for Eye Protection During Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 13262
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-06

CONDITIONS: Eyelid Erythema

STUDY DESIGN:
Intervention Model Description: The investigators will perform a prospective, double-blind, randomized controlled trial. The co-investigator will ask the study subject to close his or her eyes and will take a photograph of the eyelids as a baseline assessment. Then, the co-investigator will apply the Transpore® on one eye and the TegadermTM on the other eye according to the randomization schema. The exact time of application will be documented. At the end of the surgery, the co-investigator will remove the Transpore® and TegadermTM. She will then take another photograph of the eyelids and document the time. The Cloud storage folder containing the photographs will be shared with the dermatologists who will evaluate the degree of erythema.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tegaderm Left (Experimental): After general anesthesia is administered, Tegaderm will be placed on the left eye and Transpore will be placed on the right eye
  Interventions: Device: Tegaderm Eye Tape
- Transpore Right (Experimental): After general anesthesia is administered, Transpore will be placed on the right eye and Tegaderm will be placed on the left eye.
  Interventions: Device: Transpore Eye Tape

INTERVENTIONS:
Device: Tegaderm Eye Tape — Eye tape to protect the eye from corneal abrasions during surgery.
  Arms: Tegaderm Left
Device: Transpore Eye Tape — Eye tape to protect the eye from corneal abrasions during surgery.
  Arms: Transpore Right

SUMMARY:
The purpose of this study is to compare the rate of eyelid erythema after anesthesia with the use of TegadermTM vs. the Transpore®. Our null hypothesis is that the rate of erythema will be similar between the two groups given there is no evidence currently to suggest otherwise

DETAILED DESCRIPTION:
At Tufts Medical Center, a variety of adhesive tapes are used to shut the eyes during anesthesia, including 3MTM TegadermTM and the Sharn Anesthesia Transpore®, with no preference for one or the other. While all of these products decrease the risk of corneal abrasion, none of these products have been shown to be superior to the others in terms of eyelid irritation. According to Sharn Anesthesia, "The [Transpore®] adhesive is light enough to reduce damage to the outer eye" (3). However, there is no scientific evidence to support this claim. All the investigators know is that the Transpore is coated with a medical grade, pressure-sensitive acrylic adhesive and that there are no phthalates, it is latex free and silicone free.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Surgeries scheduled for anesthesia of any duration

Exclusion Criteria:

* Any patient that does not consent
* Any patient who has:
* Pre-existing eyelid erythema or other eyelid trauma
* Eyelid piercings
* Any surgery on the head, brain, neck, teeth, mouth, eyes, or face
* Surgery in the prone position
* Patients less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
The proportion of eyelids with erythema at the end of surgery after removal of Tegaderm vs. Transpore | Immediately after tape removal
  Degree of erythema seen in the photo taken of the eyelid immediately after the tape is removed after surgery

SECONDARY OUTCOMES:
Epidermal Change | Immediately after tape removal
  Any epidermal changes seen on the eyelid
Edema | Immediately after tape removal
  Edema seen after eye tape removal

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share the individual participant data. The individual patient records will be kept secure in an office setting.

REFERENCES:
- [Background] Cucchiara RF, Black S. Corneal abrasion during anesthesia and surgery. Anesthesiology. 1988 Dec;69(6):978-9. doi: 10.1097/00000542-198812000-00034. No abstract available. PMID 3195772
- [Background] Zeng LA, Lie SA, Chong SY. Comparison of Medical Adhesive Tapes in Patients at Risk of Facial Skin Trauma under Anesthesia. Anesthesiol Res Pract. 2016;2016:4878246. doi: 10.1155/2016/4878246. Epub 2016 Jun 12. PMID 27382368